CLINICAL TRIAL: NCT00796328
Title: Up-down Determination of the ED90 of the Initial Rate of Infusion of Phenylephrine for the Prophylaxis of Spinal Induced Hypotension in Parturients Undergoing Cesarean Delivery
Brief Title: Up-Down Determination of the ED90 of Phenylephrine for Hypotension Prophylaxis in Cesarean Delivery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Results Invalid, study closed, analysis cannot proceed.
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IWK-4462-2008
Record Dates: First submitted 2008-11-19; First posted 2008-11-24 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Spinal Induced Hypotension in Cesarean Delivery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Phenylephrine infusion

INTERVENTIONS:
Drug: Phenylephrine infusion — Up-down, biased coin design

SUMMARY:
This study is designed to determine the ED90 for an infusion of phenylephrine to prevent spinal induced low blood pressure in parturients presenting for an elective cesarean delivery. The up-down methodology (UDM) is commonly used study method to determine the dose of a drug that causes the desired effect in over 90% of the subjects to whom it given. For example: the investigators want to know what is the best dose of phenylephrine (from a range of commonly used doses) to prevent a drop in blood pressure during cesarean delivery ninety times out of one hundred when it is given at that dose. The ED90 is the effective dose at which 90% of subjects will have a "positive" response to a phenylephrine infusion, i.e. no drop in blood pressure. The investigators hypothesize that the ED90 will be between 40 - 60 mcg/min.

The primary outcome measure is the ED90 for phenylephrine infusions that prevents a drop in blood pressure in women undergoing cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent cesarean delivery with planned spinal anesthesia (i.e. elective planned cesarean delivery for malposition, patient choice, cervical pelvic disproportion, previous cesarean delivery and other diagnosis that require a predetermined cesarean delivery)
2. American Society of Anesthesia physical status class I & II (ASA I - Healthy, ASA II - mild and controlled systemic disease, eg. controlled essential hypertension)
3. Age ≥ 18 years (Standard within the obstetrical literature)
4. Term gestational age
5. English-speaking

Exclusion Criteria:

1. Morbid Obesity (Body Mass Index ≥ 45 kg/m2) (Morbidly obese parturients require a dose of local anesthetic less than the standardized dose in this study, typically have an exaggerated response to vasopressors, and the blood pressure cuff occasionally needs to be replaced by an intra-arterial catheter due to limitations in size)
2. Height < 5'0" (Women < 5'0" are likely to require a dose of local anesthetic less than the standardized dose in this study)
3. Laboring women
4. Urgent or emergency cesarean delivery
5. Hypertensive disease of pregnancy
6. Severe maternal cardiac disease
7. Subjects on monoamine oxidase inhibitors (MAOI's) or tricyclic antidepressants
8. Fetal anomalies or intrauterine fetal death
9. Failed spinal anesthesia
10. Subject enrollment in another study involving a study medication within 30 days of CD
11. Any other physical or psychiatric condition which may impair their ability to cooperate with study data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six subjects were withdrawn from the study
Groups:
- Phenylephrine Infusion: Phenylephrine infusion : Up-down, biased coin design
Period: Overall Study
Arm/Group | Phenylephrine Infusion
Started | 46
Completed | 40
Not Completed | 6
Not completed — experienced hypotension requiring tx | 6

BASELINE CHARACTERISTICS:
Arm/Group | Phenylephrine Infusion
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Effective Dose of Phenylephrine at Which 90% of Subjects Have no Spinal Induced Hypotension
Description: The effective dose at which 90% of subjects will have a "positive" response to a phenylephrine infusion, i.e. no spinal induced hypotension. We hypothesize that the ED90 will be between 40 - 60 mcg/min.
Time Frame: Spinal administration until delivery
Measure: Number; unit: dose of phenylephrine
Arm/Group | Phenylephrine Infusion
Number analyzed (Participants) | 40
dose of phenylephrine | NA — An error in the up-down sequencing was discovered. The subsequent participants would have allocated to a dose incorrectly as per the biased coin design. The results are invalid.

ADVERSE EVENTS:
Arm/Group | Phenylephrine Infusion
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No